CLINICAL TRIAL: NCT03617900
Title: EFFICACY OF GINGER EXTRACT ON PAIN RELIEF FOR FIRST NORMAL POSTPARTUM WOMEN
Brief Title: Efficacy of Ginger Extract (Compare Between the Ginger Preparation of Ancient Concept of Thai Traditional Practitioner, Standard Drug and Placebo) by Using Pain Score to Evaluate After Pain of Three Groups of First Normal Postpartum Women.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Naphatsaran Roekruangrit, Principle investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Thammasat University
Record Dates: First submitted 2018-06-11; First posted 2018-08-07 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Postpartum Disorder
Keywords: ginger extract; pain relief; postpartum women
MeSH Terms: conditions — Puerperal Disorders | interventions — ginger extract; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule; Drug: Paracetamol
- Ginger (Experimental)
  Interventions: Drug: Ginger; Drug: Paracetamol
- Paracetamol (Active Comparator)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Ginger — Ginger extract is contains 100 mg/capsules. Use 2 capsules 3 times/day
  Arms: Ginger
Drug: Placebo oral capsule — Lactose monohydrate 400 mg/capsules
  Arms: Placebo
Drug: Paracetamol — 500 mg paracetamol. use in need

SUMMARY:
Introduction A common problem in women after childbirth is bleeding (5-8 percent). This is one of the leading causes of maternal death in Thailand. The incidence of postpartum hemorrhage is approximately 1-2 percent of the births. A second problem is infection after birth which is a leading cause of illness and death of the mother. Incidence of infection after childbirth is 1-2 percent of women in developed countries and 5-10 percent of postpartum women overall. Staphylococcus aureus bacterium is found in the reproductive system of 5-9 percent of women. Perineal wound infections cause perineal pain. Thirdly is the problem of insufficient milk in foreign countries, mothers breastfeeding for less than 12 months total 94.7 percent. The fourth problem is difficult urination after vaginal delivery or 6 hours after removing the catheter in surgical cases. It is a common and important problem from 1.7 to 17.9 percent. The above problem causes infection and inflammation pain.

The first 24 hours after birth to 6 weeks physical and physiological changes of maternal organs and systems occurs such as the decline in hormone levels. This includes human placental lactogen (HPL), human chorionic somatomammotropin (HCS), human chorionic gonadotropin (HCG), estrogen, progesterone, prolactin, follicular stimulating hormones, luteinizing hormones. There is also blood loss. The clinical difficulties found in the postpartum period include after pain, perineal pain, breast engorgement, puerperal diuresis, weight loss, fever, pain and discomfort after birth. And the pain decreases or is lost in 3 days after birth.

The original gate-control theory proposed that there is a physiological within the substantia gelatinosa of the spinal cord's dorsal horn grey matter. It is suggested that sensory signals can only pass through the cells in the substantia gelatinosa when the gate is open. When the gate is closed, sensory information is blocked, and this forms the basis of a kind of physiological pain relief.

In relation to the 4 basic life elements of earth, water, wind and fire, the maternal body is lacking wind. This causes the fire to also decrease and the element of pain results. It becomes important to restore balance by stimulating blood circulation and herbal treatment is desirable to help the fire of the blood to speed the element of wind through the body.

Thai Traditional Medicine is used to treat the pain of mothers after childbirth. Because of in balance of mind fire in the body. By this reason, the balance of fire and wind increase to spread the circulatory system. Medicinal plants can increase the element of fire and the wind. Also, in Thai Traditional Medicine concept, pain reduction for postpartum mothers includes regular massage, herbal steam, herbal breast compress, Tub Mhor Kluer, eating heat-producing food. In the Thai Traditional Medicine manuscript, Kam-pee Mahachotharat there are 85 remedies for blood treatment therapy and especially, 44 contain ginger. Representing 51.76 percent of then.

Ginger has been included in the National Essential Medicines Catalogue 2554. Medication to relieve heartburn, bloating and distension, is documented and prevention and relief of nausea and vomiting due to motion sickness, seasickness. Or after surgery, are all included.

DETAILED DESCRIPTION:
1.2 Objectives

1.2.1 Primary Objective To compare the efficacy of ginger extract on pain relief at the following anatomical locations. Uterus, episiotomy and breast.

1.2.2 Secondary Objectives 1.2.2.1 To study the biological activity and stability of ginger extract. 1.2.2.2 To compare pain scores by using ginger extract for first normal postpartum women.

1.3 Benefit of Output 1.3.1 Knowledge on standard and the stability of ginger extract. 1.3.2 Knowledge on the effectiveness of ginger extract on pain relief for first normal postpartum women.

1.3.3 Knowledge on clinical research of pain relief for first normal postpartum women in the next big group volunteers.

1.3.4 Agencies involved in the field of conventional medicine and Thai Traditional Medicine may use results for study, further research and development of new drugs.

1.4 Operational Definition 1.4.1 Efficacy of ginger extract referred to changes result from receive ginger extract.

1.4.2 Pain referred to IASP (International Association for the Study of Pain) pain that persists beyond normal healing time p>24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Being 20-34 years of age.
3. First normal, healthy showing no symptoms of disorder. No history of toxemia of pregnancy, liver disease, kidney disease and gastrointestinal bleeding during pregnancy or after participating in a research project.
4. Healthy pregnant women.
5. No postpartum hemorrhage.
6. Agrees to consent form.
7. No need to take medication regularly.
8. No smoking, no drinking alcohol during pregnancy.

Exclusion Criteria:

1. Unable to travel conveniently.
2. Allergic to modern medicine or herbal remedies.
3. Have a gallstone problem.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scores on the numeric rating scale at 3 days | 2 hours after delivery time and be continued every 6 hours for 3 days.
  measurement tool is numeric rating scale: NRS. Score from 0 to 10. Inclusion criteria start at Pain was classified as Mild (1-3), Moderate (4-6), and Severe (7-10).

CONTACTS AND LOCATIONS:
Overall Officials: Preecha Wanichsetakul, M.D., Study Chair — Thammasat University; Arunporn Itharat, PH.D., Study Chair — Thammasat University
Locations (1):
- Naphatsaran Roekruangrit, Pathum Thani, Thailand

REFERENCES:
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388